CLINICAL TRIAL: NCT04757701
Title: The Role of Dentists in HPV Vaccination: Building the Infrastructure Between Co-located Dental Practices and Federally Qualified Health Centers to Facilitate HPV Vaccination Uptake
Brief Title: The Role of Dentists in Human Papillomavirus Vaccination
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: East Carolina University (Other)
Responsible Party: Sponsor
Other Study IDs: 60585
Record Dates: First submitted 2021-01-27; First posted 2021-02-17 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-03

CONDITIONS: HPV
MeSH Terms: interventions — Interviews as Topic; Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General dentists and dental hygienists in North Carolina: This objective will be met by administering a quantitative survey to active and licensed NC dentists and dental hygienists.
  Interventions: Other: Social Behavioral surveys, interviews, and focus groups
- Directors of Service-Learning Centers and their partnering FQHCs: This objective will be met by conducting qualitative assessments with ECU's SoDM's CSLCs and their partnering community clinic/FQHCs. The investigators will interview the Directors of the eight existing CSLCs and focus groups with clinical staff at each CSLC. In collaboration with the Directors of the CSLCs, the investigators will identify key stakeholders in the co-located/partnering medical clinics, and conduct interviews with the administrators and focus groups with medical clinic staff.
  Interventions: Other: Social Behavioral surveys, interviews, and focus groups

INTERVENTIONS:
Other: Social Behavioral surveys, interviews, and focus groups — Surveys with dentists/hygienists, interviews/focus groups with service learning center directors and key staff at federally qualified health centers.

SUMMARY:
This project involves the research into understanding the functioning of co-located/partnering dental practices and federally qualified health centers/community health clinics in North Carolina and how dental health providers may play a role in facilitating HPV vaccination uptake for under-vaccinated populations in these co-located/partnering sites.

DETAILED DESCRIPTION:
Objective 1): To assess HPV-related Oropharyngeal Cancer (OPC) knowledge, perceptions, practices and barriers of general dentists and dental hygienists in North Carolina (NC).

Objective 2): To understand key infrastructure elements and policies, as well as HPV prevention strategies in place at East Carolina University School of Dental Medicine Community Service-Learning Centers (CSLCs) and their partnering Community Health Clinics/Federally Qualified Health Clinics (FQHCs).

Objective 3): Develop and assess the feasibility of a model for collaborative and effective HPV prevention strategies between dental practices (CSLCs) and co-located Community Health Clinics (FQHCs).

Hypotheses:

H1. It is hypothesized that HPV OPC knowledge, perceptions, and practices will be informed by level of HPV health literacy; where higher levels of HPV health literacy will correlate with higher levels of HPV prevention practices (i.e., oral cancer screening, education on HPV risk behaviors, HPV vaccine recommendation). The investigators expect to find gaps in one or more of the surveyed areas (knowledge, attitudes, societal norms, perceived behavior control, and current prevention practices) among dentists and dental hygienists. Last, the investigators expect to find barriers to HPV prevention practices among our sample.

H2: It is hypothesized that there will be key infrastructure elements and policies identified through interviews that will both inhibit and facilitate the navigation of patients for HPV vaccination between dental clinics (CSLCs) and partnering health clinics (community clinics/FQHCs). The investigators also expect to find a variation of HPV prevention strategies currently being employed at CSLCs and partnering community clinic/FQHCs.

H3: It is hypothesized that the investigators will employ the data identified in Objectives 1 and 2 to develop a feasible model for collaborative and effective HPV prevention between dental clinics (CSLCs) and health clinics (FQHCs). Specifically, the investigators will address barriers identified in Objective 2 and capitalize on the facilitators identified to develop a model of HPV prevention care and navigation between dental clinics (CSLCs) and health clinics (FQHCs). This model can then be evaluated for effectiveness and serve as a model for replication in other rural and under-resourced settings.

ELIGIBILITY:
Inclusion Criteria:

* licensed and active dentists and hygienists in NC
* Directors/administrators of the identified CSLCs (n=8) and partnering FQHCs/Community clinics (n=8)

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Objective 1 Population: licensed and active dentists in NC, and licensed and active dental hygienists.
  Objective 2 Population: Current locations of the eight CSLCs include Ahoskie (Hertford County), Elizabeth City (Pasquotank County), Lillington (Harnett County), Sylva (Jackson County), Lumberton (Robeson County), Davidson (Davidson County), Spruce Pine (Mitchell County), and Brunswick (Brunswick County). The investigators will also identify key stakeholders from partnering FQHC/Community Health Clinics to include in qualitative interviews.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Quantitative measurements of the following variables: HPV-related Oropharyngeal Cancer knowledge, perceptions, practices and barriers as measured by a dental questionnaire to be developed by study team | Year 1
  HPV-related Oropharyngeal Cancer (OPC) knowledge, perceptions, practices and barriers of general dentists and dental hygienists in North Carolina. The dental questionnaire will be developed by study investigators and will use validated survey items, and will be piloted, and tested for readability, reliability, and validity by the research team.
  Use of the survey is a quantitative technique; the resulting validated data of the dental questionnaire suggests predictable outcomes.
Qualitative open ended statements will be assessed through qualitative interviews and focus groups which will generate a list of key infrastructure elements and policies, and HPV prevention strategies | Year 2
  Through qualitative assessments of interviews and focus groups with East Carolina University School of Dental Medicine Community Service-Learning Centers and their partnering community clinic/FQHCs, study investigators will develop a list of key infrastructure elements and policies, as well as HPV prevention strategies in place at East Carolina University School of Dental Medicine Community Service-Learning Centers and their partnering Community Health Clinics/Federally Qualified Health Clinics.
  Use of qualitative assessments with comparative reviews of EMR data suggests a validation schema to predict infrastructure needs and outcomes.
Study investigators will also conduct a review of the Electronic Medical Records of both dental and partnering medical clinic to assess how HPV-related screenings, vaccinations, and malignancies are reported | Year 2
  Study investigators will also conduct a review of the Electronic Medical Records of both dental and partnering medical clinic to assess how HPV-related screenings, vaccinations, and malignancies are reported

CONTACTS AND LOCATIONS:
Overall Officials: Essie Torres, PhD, Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Winterville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No